CLINICAL TRIAL: NCT05766254
Title: Identify the Optimal TMS Target to Modulate Midcingulate Reward Activity in Smokers
Brief Title: Identify the Optimal TMS Target to Modulate Reward Activity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Travis Baker, PhD, Assistant Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro2022000444
Record Dates: First submitted 2023-02-21; First posted 2023-03-13 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Nicotine Use Disorder
Keywords: transcranial magnetic stimulation; reward processing; EEG; neuroimaging
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single (Participant) Participants will be blinded as to TMS condition (active or sham)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active TMS (Experimental): Participants in the active condition will receive repetitive TMS (rTMS), delivered at 110% of participants' resting motor threshold at 10 Hz continuously over the predefined prefrontal target for a total of 1000 pulses. Within each of the two TMS sessions, two targets will be stimulated.
  Interventions: Device: Active 10-Hz TMS to the DLPFC
- Sham TMS (Sham Comparator): Identical parameters will be applied to the SHAM group with the exception that the TMS coil will be flipped 180º to mimic auditory stimulation.
  Interventions: Device: Sham TMS-DLPFC

INTERVENTIONS:
Device: Active 10-Hz TMS to the DLPFC — The active group will receive 10hz TMS stimulation. Participants in the active stimulation group will receive10-Hz TMS to left DLPFC. The LDLPFC will be based on 4 targeting neuroimaging methods (cortical thickness, fMRI, diffusion imaging, functional connectivity). TMS will be delivered using a robotic neuronavigation system (Smartmove, ANT). Stimulation intensity will be standardized at 110% of RMT and adjusted to the skull to cortical surface based on e-field calculations (simnibs). Stimulation will be delivered to the L-DLPFC using a active/placebo figure-8 coil and a magventure TMS device.
  Arms: Active TMS
Device: Sham TMS-DLPFC — The parameters in the active arms will be as above with the internal randomization of the device internally switching to sham in a blinded fashion.
  Arms: Sham TMS

SUMMARY:
Our primary goal will be to identify the optimal prefrontal-cingulate target by systematically measuring the efficacy of various image-based targeting techniques to increase the reward positivity using the 10-Hz TMS protocol in dependent smokers. Our secondary objective will be to measure the targets' effectiveness to increase decision-making capacity using the probabilistic selection task (PST). Our third objective will be to specifically assess whether the TMS targets has a differential impact on state levels of craving relative to baseline (Tobacco Craving Questionnaire [TCQ]. We plan to accomplish these three objectives using a randomized, controlled experiment involving 3 sessions.

DETAILED DESCRIPTION:
The design is primarily a randomized control-trial design (3 sessions), comparing the effects 10-Hz rTMS applied to four prefrontal TMS targets based on fMRI, cortical thickness (CT), diffusion-weighted imaging (DWI) and resting state functional connectivity (RSFC) on reward processing across two groups of smokers - Active TMS group and Sham TMS group. For Session A, participants will be scanned using a 3 Tesla MRI system and will receive a structural (T1), fMRI, DWI, and resting-state FC scan. Following Session A, all participants will be asked to complete two Ri-TMS sessions within two weeks and will be instructed to abstain from smoking for 4 hours before the start of each scheduled session. Session B and C: Distinct prefrontal target regions will be identified for each subject based on CT, fMRI, DWI, and RSFC data. At the start of Session B, a target will be randomly assigned to each subject using a random permuted block method. For Sessions B and C, participants will be asked to provide their consent, CO levels, and complete the craving questionnaire (TCQ). At the start of Session B, participants will be fitted with an EEG cap and engage in a virtual T-maze feedback task. The task will be divided into two blocks (200 trials per block: 10 minutes per block). At the start of Block 1, the robotic arm will position the TMS coil <1 cm over Target 1. Next, 50 rTMS pulses will be delivered at 110% of participants' rMT at 10- Hz continuously over Target 1 immediately before every 10 trials of the T-maze (5 seconds of TMS, 30 seconds of task). A total of 1000 pulses will be delivered to Target 1 and 200 T-maze trials completed (duration 10-15 minutes). Immediately after, subjects will be asked to complete a probabilistic selection task (PST) to measure post-stimulation effects on decision-making performance (duration, 15 minutes). Following the completion of the PST, subjects will be given a 5 minute rest-break and participants will be asked to fill out the TCQ. At the start of Block 2, the robotic arm will position the TMS coil <1 cm over Target 2, and 50 rTMS pulses will be delivered immediately before every 10 trials of the T-maze task. A total of 1000 pulses will be delivered to Target 2 and 200 T-maze trials completed (duration 10 minutes). Following Target 2 stimulation, subjects will be asked to complete the PST (duration, 15 minutes) and asked to fill out the TCQ. At the end of the Session B, participants will be scheduled to return to the laboratory to complete Session C on a separate day. An identical protocol will be applied to Session C with the exception that TMS pulses will be deliver to Target 3 and Target 4.

ELIGIBILITY:
Inclusion Criteria:

1. Nicotine dependent individuals (according to the Alcohol, Smoking and Substance Involvement Screening Test nicotine dependence score).
2. Be between the ages of 18 and 55 years old.
3. Not received substance abuse treatment within the previous 30 days.
4. Be in stable mental and physical health.
5. If female, test non-pregnant.
6. No evidence of focal or diffuse brain lesion on MRI.
7. Be willing to provide informed consent.
8. Be able to comply with protocol requirements and likely to complete all study procedures.

Exclusion Criteria:

1. Contraindication to MRI (e.g., presence of metal in the skull, orbits or intracranial cavity, claustrophobia).
2. Contraindication to rTMS (history of neurological disorder or seizure, increased intracranial pressure, brain surgery, or head trauma with loss of consciousness for > 15 minutes, implanted electronic device, metal in the head, or pregnancy).
3. History of autoimmune, endocrine, viral, or vascular disorder affecting the brain.
4. History or MRI evidence of neurological disorder that would lead to local or diffuse brain lesions or significant physical impairment.
5. Life time history of mental disorders such as: Bipolar Affective disorder (BPAD), Schizophrenia, Post-traumatic Stress disorder (PTSD) or Dementia or Major Depression.
6. uninterruptable central nervous system medication

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-03-24 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Event-related Brain Potential: Reward Positivity | Day 0 (day of testing)
  The reward positivity is an event-related brain potential (ERP) sensitive to reward feedback. The reward positivity will be measured during the T-maze task, where participants will receive feedback (Reward, No-reward) following choices. ERPs will be created for each electrode and participant by averaging the single-trial EEG according to feedback type (Reward, No-reward). The reward positivity will be evaluated by subtracting the Reward feedback ERPs from the corresponding No-reward feedback ERPs. The size of the reward positivity will then be determined by identifying the maximum absolute amplitude of the difference wave within a 200-to 400-msec window after feedback onset and evaluated along electrodes Fz, FCz, and Cz. The reward positivity will be measured for each proposed DLPFC target across active and sham groups of dependent smokers. The reward positivity will be used to measure the efficacy of the DLPFC target to modulate reward activity.

SECONDARY OUTCOMES:
Approach Learning | Day 0 (day of testing)
  Approach learning will be measured using a Probabilistic Selection task (PST), in which subjects are shown pairs of arbitrary stimuli and must learn by trial-and-error to select one of each pair. During an initial learning phase participants are exposed to three pairs of stimuli, each of the three pairs is rewarded on 80%, 70%, and 60% of the trials. Subjects learn by feedback that some stimuli are associated with more positive feedback (Approach) and that some stimuli are associated with more negative feedback (Avoidance). To determine whether subjects learn more from positive (approach) or negative (avoidance) feedback, during a subsequent testing phase they are required to choose between novel stimulus pairs. Approach learning (accuracy and reaction time) for each proposed DLPFC target across active and sham groups will be measured during the testing phase. Avoidance learning performance will be used to measure the efficacy of the DLPFC target to modulate decision making.
Avoidance Learning | Day 0 (day of testing)
  Avoidance learning will be measured using a Probabilistic Selection task (PST), in which subjects are shown pairs of arbitrary stimuli and must learn by trial-and-error to select one of each pair. During an initial learning phase participants are exposed to three pairs of stimuli, each of the three pairs is rewarded on 80%, 70%, and 60% of the trials. Subjects learn by feedback that some stimuli are associated with more positive feedback (Approach) and that some stimuli are associated with more negative feedback (Avoidance). To determine whether subjects learn more from positive (approach) or negative (avoidance) feedback, during a subsequent testing phase they are required to choose between novel stimulus pairs. Avoidance learning (accuracy and reaction time) for each proposed DLPFC target across active and sham groups will be measured during the testing phase. Avoidance learning performance will be used to measure the efficacy of the DLPFC target to modulate decision making.
Nicotine Craving | Day 0 (day of testing - before and after TMS)
  The level of craving will be assessed in dependent smokers using the short version of the Tobacco Craving Questionnaire (TCQ), a 12-item scale that assesses state levels of craving. TCQ will be measured at the start of each session, and following each Block of TMS (once for each DLPFC target). We will compared the TCQ score from pre-TMS (start of session) to post-TMS.

CONTACTS AND LOCATIONS:
Overall Officials: Travis E Lalta, PhD, Principal Investigator — Rutgers University
Locations (1):
- Rutgers University - Newark, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
Data may be uploaded to an open source framework. All data will be deidentified.